CLINICAL TRIAL: NCT07009561
Title: Comparison of Cortical Excitability and Typing Performance Across Action Observation, Motor Execution, and Control Conditions
Brief Title: Cortical Excitability and Typing Performance After Action Observation and Motor Execution
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sharjah (Other)
Responsible Party: Principal Investigator, Meeyoung Kim, Assistant professor, University of Sharjah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: TMStyping
Record Dates: First submitted 2025-05-29; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Young Adults
Keywords: Transcranial magnetic stimulation; Cortical excitability; Action observation; Motor execution; Typing

STUDY DESIGN:
Intervention Model Description: This study will be a prospective, double-blinded, parallel, randomized controlled trial. A total of 60 participants will be randomly assigned into three groups: Motor Execution (ME), Action Observation (AO), and Control. Each group will consist of 20 participants. Interventions will include a 3-minute typing task (ME), a 3-minute observation video (AO), or no task (Control). All participants will undergo pre- and post-intervention typing and TMS assessments.
Who Masked: Participant, Outcomes Assessor
Masking Description: This will be a double-blinded randomized controlled trial in which participants will be unaware of their group allocation or the purpose of the intervention they receive. Outcome assessors and data analysts will also be blinded to the group assignments. To ensure assessor blinding, TMS and typing data will be coded and analyzed by an independent researcher who is not involved in intervention delivery or participant interaction. The interventions (ME, AO, Control) will be conducted in a standardized format, minimizing interaction and disclosure that could bias results.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ME (Experimental): Participants will undergo pre and post assessments. Each assessment include Transcranial Magnetic Stimulation (TMS) and typing performance tests.
  Pre-assessment will be conducted in the first visit.
  In the second visit, Motor Execution (ME) group will perform a 3-minute typing task using both hands in a standardized posture. The typing task will consist of custom-designed text that emphasizes use of the index finger, matching the target muscle for TMS.
  Participants will then undergo post-assessment as same as the pre-assessment within 15 minutes after completing the typing task.
  There will be time window more than 48 hours between visits.
  Interventions: Behavioral: Motor Execution Typing Task
- AO (Experimental): Participants will undergo pre and post assessments. Each assessment include Transcranial Magnetic Stimulation (TMS) and typing performance tests.
  Pre-assessment will be conducted in the first visit.
  During the second visit, participants in the Action Observation (AO) group will observe a 3-minute first-person point-of-view video of a person typing the same standardized text used in the ME group. The video will emphasize index finger movement on a QWERTY keyboard.
  Participants will then undergo post-assessment as same as the pre-assessment within 15 minutes after watching the typing video.
  There will be time window more than 48 hours between visits.
  Interventions: Behavioral: Action Observation of Typing Task
- Control (No Intervention): Participants in the Control group will not receive any intervention between the pre- and post-assessments.
  They will undergo the same assessments as the other groups to allow comparison of changes in cortical excitability and typing performance.
  There will be time window more than 48 hours between visits.

INTERVENTIONS:
Behavioral: Motor Execution Typing Task — Participants will perform a 3-minute typing task using custom-designed text that emphasizes index finger use. This task is designed to actively engage the motor cortex and will be administered in a controlled environment using standard posture and equipment. The task aims to elicit changes in cortical excitability, which will be measured pre- and post-intervention using TMS.
  Arms: ME
Behavioral: Action Observation of Typing Task — Participants will observe a 3-minute first-person video of an individual typing the standardized text. The video is designed to activate mirror neuron systems through visual engagement with a familiar motor task. It will be shown once in a controlled setting, and post-assessment of cortical excitability will follow immediately after.
  Arms: AO

SUMMARY:
Goal:

This study will aim to investigate the effects of different motor stimulation strategies-motor execution (ME) and action observation (AO)-on cortical excitability and typing performance in healthy individuals.

Recruitment:

A total of 60 healthy university students will be recruited and randomly assigned into three groups:

Motor Execution group (n=20) Action Observation group (n=20) Control group (n=20)

Evaluation Tools:

Transcranial Magnetic Stimulation (TMS) using DEYMED DuoMAG XT will be used to measure Resting Motor Threshold (RMT), Motor Evoked Potential (MEP) Amplitude, and MEP Latency of the First Dorsal Interosseous (FDI) muscle.

Online Typing Test will be used to assess typing speed (words per minute) and accuracy (percentage of correct characters).

Intervention:

The ME group will perform a 3-minute typing task. The AO group will observe a 3-minute first-person video of typing. The Control group will not receive any intervention between assessments.

All participants will undergo TMS and typing assessments twice, once before and once after the intervention.

DETAILED DESCRIPTION:
This study will be designed as a randomized controlled trial to compare the effects of motor execution (ME) and action observation (AO) on cortical excitability and fine motor performance, using typing as the target motor task.

A total of 60 healthy university students will be recruited from the University of Sharjah through convenience sampling. Participants will be screened based on inclusion and exclusion criteria and will provide informed consent prior to enrollment. Eligible participants will then be randomly assigned into three groups (ME, AO, and Control), with stratification based on baseline typing proficiency to ensure balanced motor skill levels across groups.

All participants will undergo a pre-assessment session that will include a 3-minute typing task focused on the index finger and TMS testing targeting the First Dorsal Interosseous (FDI) muscle. TMS measures will include Resting Motor Threshold (RMT), MEP Amplitude, and MEP Latency.

During the intervention phase:

The ME group will perform the typing task for 3 minutes. The AO group will watch a 3-minute point-of-view video of the same typing task. The Control group will receive no intervention and will simply wait between the assessments.

After the intervention, participants in all groups will repeat the same typing task and TMS assessments in the post-assessment phase.

Typing performance will be evaluated using an online typing platform, capturing typing speed (words per minute) and accuracy (percentage of correct characters). TMS data will be collected using the DEYMED DuoMAG XT with consistent coil placement and stimulation parameters. Five reproducible MEPs will be recorded per participant per session to ensure reliability.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 26 years
* Healthy university students with no known neurological, psychiatric, or musculoskeletal conditions
* Intact motor functioning of the upper limbs
* Basic typing proficiency using a 10-finger typing method
* Ability to understand study procedures and provide informed consent

Exclusion Criteria:

* Typing speed less than 16 words per minute
* Use of hunt-and-peck or single-finger typing style
* History of seizures or epilepsy
* Current use of neuroactive medications
* Presence of metallic implants in the head or upper body
* Any contraindications to Transcranial Magnetic Stimulation (TMS)
* Left-handed individuals using non-standard typing techniques (unless provided with adapted materials)

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Change in Resting Motor Threshold (RMT) | Pre-intervention (Day 1) and Post-intervention (within 15 minutes after intervention on Day 2, between 48 hours to a 3-week window)
  Resting Motor Threshold (RMT) will be measured using Transcranial Magnetic Stimulation (TMS) targeting the First Dorsal Interosseous (FDI) muscle. RMT is defined as the minimum stimulation intensity required to evoke a measurable motor evoked potential (MEP) of ≥50 µV in at least 5 out of 10 trials.
Change in MEP Latency and Amplitude | Pre-intervention (Day 1) and Post-intervention (within 15 minutes after intervention on Day 2, between 48 hours to a 3-week window)
  Motor Evoked Potential (MEP) latency (in milliseconds) and amplitude (in µV) will be assessed using TMS. These measures reflect neural conduction time and the magnitude of cortical response, respectively.
Change in Typing Speed (Words Per Minute) | Pre-intervention (Day 1) and Post-intervention (within 15 minutes after intervention on Day 2, between 48 hours to a 3-week window)
  Typing speed will be measured using a standardized online typing platform, expressed in words per minute (WPM). Participants will complete a 3-minute typing task using custom text emphasizing index finger usage.
Change in Typing Accuracy | Pre-intervention (Day 1) and Post-intervention (within 15 minutes after intervention on Day 2, between 48 hours to a 3-week window)
  Typing accuracy will be recorded as the percentage of correctly typed characters during a 3-minute standardized typing task using an online platform.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Sharjah, University City, Emirate of Sharjah, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) collected during the study will be made available to qualified researchers upon reasonable request. Data will be shared for the purpose of academic research and meta-analyses related to motor learning, neuroplasticity, and rehabilitation.
Supporting Information: Study Protocol, SAP
Time Frame: After 6 months of completing a study and available for one year
Access Criteria: Access will be granted to academic researchers affiliated with recognized institutions for non-commercial research purposes only. Approved researchers must sign a data use agreement, ensuring the data will be used solely for the approved purpose, will not be re-identified, and will be securely stored.
  Priority will be given to proposals that aim to expand scientific knowledge on motor learning, neuroplasticity, TMS, or physiotherapy interventions.

REFERENCES:
- [Background] Bhattacharya A, Mrudula K, Sreepada SS, Sathyaprabha TN, Pal PK, Chen R, Udupa K. An Overview of Noninvasive Brain Stimulation: Basic Principles and Clinical Applications. Can J Neurol Sci. 2022 Jul;49(4):479-492. doi: 10.1017/cjn.2021.158. Epub 2021 Jul 9. PMID 34238393
- [Background] Birdsong D. Plasticity, Variability and Age in Second Language Acquisition and Bilingualism. Front Psychol. 2018 Mar 12;9:81. doi: 10.3389/fpsyg.2018.00081. eCollection 2018. PMID 29593590
- [Background] Grilc N, Valappil AC, Tillin NA, Mian OS, Wright DJ, Holmes PS, Castelli F, Bruton AM. Motor imagery drives the effects of combined action observation and motor imagery on corticospinal excitability for coordinative lower-limb actions. Sci Rep. 2024 Jun 6;14(1):13057. doi: 10.1038/s41598-024-63758-6. PMID 38844650
- [Background] Ma ZZ, Wu JJ, Hua XY, Zheng MX, Xing XX, Ma J, Li SS, Shan CL, Xu JG. Brain Function and Upper Limb Deficit in Stroke With Motor Execution and Imagery: A Cross-Sectional Functional Magnetic Resonance Imaging Study. Front Neurosci. 2022 May 19;16:806406. doi: 10.3389/fnins.2022.806406. eCollection 2022. PMID 35663563